CLINICAL TRIAL: NCT00593983
Title: Peer-Driven Intervention to Enroll Minorities/Women in HIV/AIDS Clinical Trials
Brief Title: Peer-Driven Intervention to Enroll Minorities/Women in HIV/AIDS Clinical Trials (the ACT2 Project)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ACT2; R01AI070005 (NIH)
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2012-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Peer-driven intervention
- 2 (Placebo Comparator): Control
  Interventions: Behavioral: Time-matched health education

INTERVENTIONS:
Behavioral: Peer-driven intervention — Consists of four structured intervention sessions lasting 6 hours in total, three peer education/recruitment experiences, and brief liaison contacts by an intervention facilitator during AIDS clinical trial screening
  Arms: 1
Behavioral: Time-matched health education — Health education and standard of care treatment
  Arms: 2

SUMMARY:
African Americans and Latinos are increasingly affected by HIV/AIDS in the United States. Despite the increase in the number of infections in minority populations, these individuals are not adequately represented in AIDS clinical trials (ACTs). The purpose of this study is to identify effective intervention strategies to increase the number of HIV infected racial/ethnic minorities and women who are screened for and enrolled into ACTs.

DETAILED DESCRIPTION:
According to a 2001 report by the U.S. Census Bureau, African Americans and Latinos make up 65% of all AIDS cases reported in the United States, yet they make up only 25% of the population in the United States. In addition, the number of women living with HIV/AIDS, many of whom are minorities, is rapidly increasing. ACTs are research studies designed to evaluate new therapies to fight HIV infection and prevent and treat opportunistic infections and cancers associated with AIDS. Preliminary research suggests that intensive intervention efforts are needed to improve rates of screening and to enroll more racial/ethnic minorities and women in ACTs. The purpose of this study is to identify effective intervention strategies to increase the low number of HIV infected racial/ethnic minorities and women who are screened for and enrolled into ACTs.

Each participant will be enrolled in the study for 12 months. Participants will be randomly assigned to either the intervention or control arm. Initial "seed" participants in the intervention arm will complete a peer-driven intervention consisting of four structured intervention sessions lasting 6 hours in total (occurring every week for 4 weeks), three peer education/recruitment experiences, and brief liaison contacts by an intervention facilitator during AIDS clinical trial screening. Participants in the control arm will complete a time-matched health education intervention lasting 6 hours. Participants in the control arm will also receive the community standard of care and be referred to their local ACT unit. Peer participants will be recruited by either a seed or through general recruitment; those recruited by an initial seed will participate in the same arm as the see d who recruited them. Study visits will occur throughout the study. Participants in the intervention arm will complete an interview at Week 30. At Weeks 8, 16 and 52, all participants will complete social impact assessments. At Weeks 16 and 52, all participants will complete follow-up visits.

ELIGIBILITY:
Inclusion Criteria for Initial Seeds:

* HIV infected
* Seen at the Betances Health Center or AIDS Service Center at least once in the last 6 months prior to study entry
* Of African-American or Latino descent
* Willing to recruit HIV infected peers
* Able to conduct research activities (e.g., speaking and writing when necessary) in English

Inclusion Criteria for Peers:

* Documented recruitment for study participation
* HIV infected
* Willing to recruit HIV infected peers
* Able to conduct research activities (e.g., speaking and writing when necessary) in English

Exclusion Criteria:

* Currently enrolled in an HIV/AIDS clinical trial
* Currently psychotic based on standard assessment (e.g., MINI, Lecrubier et al., 1997)
* Any condition that, in the opinion of the investigator, would interfere with participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2007-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Participation in screening for AIDS clinical trials to the point of determining eligibility, coded as yes/no. | within the participant's 52 week follow up period
  During interventions, participants in both arms receive contact information for local AIDS clinical trials units. Two sources of data are used to determine whether screening occurred. First, for participants screened at Beth Israel Medical Center, the study's main collaborating site, the screener notes the screening event in a participant status file. Second, during follow-up interviews at 16 and 52 weeks post-baseline, participants' screening experiences at other units are assessed. This self-reported screening is confirmed with the clinical trials units (all screening reports are verified).

SECONDARY OUTCOMES:
Enrollment into an AIDS clinical trial or HIV/AIDS biomedical research study | within the participant's 52 week follow-up period
  Two sources of data are used to determine whether enrollment occurred. First, for participants screened at Beth Israel Medical Center, the study's main collaborating site, study staff confirms participation in the trial with participants and trials units and log this in a participant status file. Second, during follow-up interviews at 16 and 52 weeks post-baseline, enrollment in studies and trials is assessed. This self-reported enrollment is confirmed with the clinical trials units (all enrollment reports are verified).

CONTACTS AND LOCATIONS:
Overall Officials: Marya Gwadz, PhD, Principal Investigator — New York University